CLINICAL TRIAL: NCT05996848
Title: Efficacy and Safety of Cagrilintide s.c. 2.4 mg in Combination With Semaglutide s.c. 2.4 mg (CagriSema s.c. 2.4 mg/2.4 mg) Once-Weekly in Chinese Participants With Overweight or Obesity
Brief Title: A Research Study to See How Well CagriSema Helps People in China With Excess Body Weight Lose Weight
Acronym: REDEFINE 6
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9838-4827; U1111-1267-4364 (Other: World Health Organization (WHO))
Record Dates: First submitted 2023-08-10; First posted 2023-08-18 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Obesity or Overweight
MeSH Terms: conditions — Obesity; Overweight | interventions — cagrilintide; semaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- CagriSema (Experimental): Participants will receive once-weekly subcutaneous (s.c) injections of 2.4 mg cagrilintide and 2.4 mg semaglutide for 44 weeks.
  Interventions: Drug: Cagrilintide; Drug: Semaglutide
- Semaglutide (Active Comparator): Participants will receive once-weekly s.c injection of 2.4 mg semaglutide for 44 weeks.
  Interventions: Drug: Semaglutide; Drug: Placebo Semaglutide
- Placebo (Placebo Comparator): Participants will receive placebo matched to cagrilintide and placebo matched to semaglutide once weekly for 44 weeks.
  Interventions: Drug: Placebo Semaglutide; Drug: Placebo Cagrilintide

INTERVENTIONS:
Drug: Cagrilintide — Participants will receive 2.4 mg cagrilintide subcutaneously.
  Arms: CagriSema
Drug: Semaglutide — Participants will receive 2.4 mg semaglutide subcutaneously.
  Arms: CagriSema; Semaglutide
Drug: Placebo Semaglutide — Participants will receive placebo matched to semaglutide subcutaneously.
  Arms: Placebo; Semaglutide
Drug: Placebo Cagrilintide — Participants will receive placebo matched to cagrilintide subcutaneously.
  Arms: Placebo

SUMMARY:
This study will look at how well the new medicine CagriSema helps people with excess body weight losing weight compared to a "dummy" medicine and a medicine called semaglutide. Participants will either get CagriSema, a dummy medicine or semaglutide. Which treatment participants get is decided by chance. Participants will take one injection once a week. The study medicine will be injected briefly with a thin needle, typically in the stomach, thighs or upper arms. The study will last for about 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age above or equal to 18 years at the time of signing informed consent

  1. Body Mass Index (BMI) greater than or equal to 30.0 kilograms per square meter (kg/m^2) or
  2. BMI greater than or equal to 27.0 kg/m^2 with the presence of at least one weight-related comorbidity including, but not limited to, type 2 diabetes mellitus, hypertension, dyslipidaemia, obstructive sleep apnoea or cardiovascular disease

For participants with Type 2 diabetes (T2D) at screening the following criteria also apply:

* Diagnosed with type 2 diabetes mellitus greater than equal to 180 days before screening
* Treatment with either lifestyle intervention, or treatment with 1-3 marketed oral antidiabetic drugs (OADs) (metformin, α-glucosidase inhibitors (AGI), glinides, sodium-glucose cotransporter 2 inhibitor (SGLT2i)), thiazolidinediones, or sulphonylureas (SUs) as a single agent or in combination) according to local label
* Treatment with oral antidiabetic drugs should be stable (same drug(s), dose and dosing frequency) for at least 60 days before screening
* Glycated Haemoglobin (HbA1c) 7 percent-10 percent (53-86 millimoles per mole [mmol/mol]) (both inclusive) as measured by the central laboratory at screening

Exclusion Criteria:

For participants without T2D at screening:

* HbA1c greater than or equal to 6.5 percent (48 mmol/mol) as measured by the central laboratory at screening
* History of type 1 or type 2 diabetes mellitus

For participants with T2D at screening:

* Clinically significant or severe hypoglycaemia within 6 months before screening or history of hypoglycaemia unawareness
* Renal impairment with estimated glomerular filtration rate (eGFR) lesser than 30 milli liter per min/1.73 meter square (mL/min/1.73 m^2), as measured by the central laboratory at screening
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a fundus examination performed within 90 days before screening or in the period between screening and randomisation. Pharmacological pupil-dilation is a requirement unless using a digital fundus photography camera specified for non-dilated examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2025-01-06 (Actual); Study Completion 2025-02-22 (Actual)

PRIMARY OUTCOMES:
CagriSema 2.4 mg/2.4 mg versus placebo: Relative change in body weight | From baseline (week 0) to end of treatment (week 44)
  Measured in percentage (%)
CagriSema 2.4 mg/2.4 mg versus placebo: Number of participants who achieve (yes/no): Body weight reduction greater than or equal to 5% | From baseline (week 0) to end of treatment (week 44)
  Measured as count of participants

SECONDARY OUTCOMES:
CagriSema 2.4 mg/2.4 mg versus placebo: Number of participants who achieve (yes/no): Body weight reduction greater than or equal to 20% | From baseline (week 0) to end of treatment (week 44)
  Measured as count of participants
CagriSema 2.4 mg/2.4 mg versus semaglutide 2.4 mg: Relative change in body weight | From baseline (week 0) to end of treatment (week 44)
  Measured in percentage (%)
CagriSema 2.4 mg/2.4 mg versus placebo: Change in waist circumference | From baseline (week 0) to end of treatment (week 44)
  Measured in centimeter (cm)
CagriSema 2.4 mg/2.4 mg versus placebo: Number of participants who achieve (yes/no): Body weight reduction greater than or equal to 10% | From baseline (week 0) to end of treatment (week 44)
  Measured as count of participants
CagriSema 2.4 mg/2.4 mg versus placebo: Number of participants who achieve (yes/no): Body weight reduction greater than or equal to 15% | From baseline (week 0) to end of treatment (week 44)
  Measured as count of participants
CagriSema 2.4 mg/2.4 mg versus semaglutide 2.4 mg: Change in waist circumference | From baseline (week 0) to end of treatment (week 44)
  Measured in centimeter (cm)
CagriSema 2.4 mg/2.4 mg versus placebo and semaglutide 2.4 mg: Change in Glycated Haemoglobin (HbA1c) | From baseline (week 0) to end of treatment (week 44)
  Measured in percentage points
CagriSema 2.4 mg/2.4 mg versus placebo and semaglutide 2.4 mg: Change in Fasting Plasma Glucose (FPG) | From baseline (week 0) to end of treatment (week 44)
  Measured as millimole per liter (mmol/L)
CagriSema 2.4 mg/2.4 mg versus placebo and semaglutide 2.4 mg: Relative change in fasting serum insulin | From baseline (week 0) to end of treatment (week 44)
  Measured in percentage (%)
CagriSema 2.4 mg/2.4 mg versus placebo and semaglutide 2.4 mg: Change in Systolic Blood Pressure (SBP) | From baseline (week 0) to end of treatment (week 44)
  Measured in millimeter of mercury (mmHg)
CagriSema 2.4 mg/2.4 mg versus placebo and semaglutide 2.4 mg: Change in Diastolic Blood Pressure (DBP) | From baseline (week 0) to end of treatment (week 44)
  Measured in millimeter of mercury (mmHg)
CagriSema 2.4 mg/2.4 mg versus placebo and semaglutide 2.4 mg: Relative change in total cholesterol | From baseline (week 0) to end of treatment (week 44)
  Measured in percentage (%)
CagriSema 2.4 mg/2.4 mg versus placebo and semaglutide 2.4 mg: Relative change in high-density lipoprotein (HDL) cholesterol | From baseline (week 0) to end of treatment (week 44)
  Measured in percentage (%)
CagriSema 2.4 mg/2.4 mg versus placebo and semaglutide 2.4 mg: Relative change in low-density lipoprotein (LDL) cholesterol | From baseline (week 0) to end of treatment (week 44)
  Measured in percentage (%)
CagriSema 2.4 mg/2.4 mg versus placebo and semaglutide 2.4 mg: Relative change in very low-density lipoprotein (VLDL) cholesterol | From baseline (week 0) to end of treatment (week 44)
  Measured in percentage (%)
CagriSema 2.4 mg/2.4 mg versus placebo and semaglutide 2.4 mg: Relative change in triglycerides | From baseline (week 0) to end of treatment (week 44)
  Measured in percentage (%)
CagriSema 2.4 mg/2.4 mg versus placebo and semaglutide 2.4 mg: Relative change in free fatty acids | From baseline (week 0) to end of treatment (week 44)
  Measured in percentage (%)
CagriSema 2.4 mg/2.4 mg versus placebo: Change in Short Form-36 Version 2.0 (SF- 36v2) Physical Functioning score | From baseline (week 0) to end of treatment (week 44)
  Measured as score points. The SF-36v2.0 is a 36-item commonly used generic clinical outcome assessment (COA) instrument measuring health-related quality of life and general health status across disease areas. SF-36v2 questionnaire measures 8 domains of functional health and well-being as well as 2 component summary scores (physical component summary and mental component summary). This endpoint assess the 'physical functioning domain'. The 0-100 scale scores from the SF-36 will be converted to norm-based scores to enable a direct interpretation in relation to the distribution of the scores in the 2009 U.S. general population. In the metric of norm-based scores, 50 and 10 correspond to the mean and standard deviation respectively. A positive change score indicates an improvement since baseline.
CagriSema 2.4 mg/2.4 mg versus placebo: Change in SF-36v2: Physical Component Summary Score | From baseline (week 0) to end of treatment (week 44)
  Measured as score points. The SF-36v2.0 is a 36-item commonly used generic COA instrument measuring health-related quality of life and general health status across disease areas. SF-36v2 questionnaire measures 8 domains of functional health and well-being as well as 2 component summary scores (physical component summary and mental component summary). This endpoint assess the 'physical component summary'. The 0-100 scale scores from the SF-36 will be converted to norm-based scores to enable a direct interpretation in relation to the distribution of the scores in the 2009 U.S. general population. In the metric of norm-based scores, 50 and 10 corresponds to the mean and standard deviation respectively. A positive change score indicates an improvement since baseline.
CagriSema 2.4 mg/2.4 mg versus placebo: Change in SF-36v2: Mental Component Summary score | From baseline (week 0) to end of treatment (week 44)
  Measured as score points. The SF-36v2.0 is a 36-item commonly used generic COA instrument measuring health-related quality of life and general health status across disease areas. SF-36v2 questionnaire measures 8 domains of functional health and well-being as well as 2 component summary scores (physical component summary and mental component summary). This endpoint assess the 'mental component summary'. The 0-100 scale scores from the SF-36 will be converted to norm-based scores to enable a direct interpretation in relation to the distribution of the scores in the 2009 U.S. general population. In the metric of norm-based scores, 50 and 10 corresponds to the mean and standard deviation respectively. A positive change score indicates an improvement since baseline.
CagriSema 2.4 mg/2.4 mg versus placebo: Change in Impact of Weight on Quality Of Life-Lite Clinical Trials Version (IWQOLLite- CT) Physical Function score | From baseline (week 0) to end of treatment (week 44)
  Measured as score points. IWQOL-Lite-CT version 3 is a 20-item COA instrument used to assess the impact of body weight changes in obesity studies on patient's physical and psychosocial functioning in three composite scores (physical function, physical and psychosocial) and a total score. This endpoint assess the 'physical function score'. The scores range between 0-100 where higher scores indicate a better quality of life. A positive change score indicates an improvement since baseline.
CagriSema 2.4 mg/2.4 mg versus placebo: Change in IWQOL-Lite-CT Total score | From baseline (week 0) to end of treatment (week 44)
  Measured as score points. IWQOL-Lite-CT version 3 is a 20-item COA instrument used to assess the impact of body weight changes in obesity studies on patient's physical and psychosocial functioning in three composite scores (physical function, physical and psychosocial) and a total score. This endpoint assess the 'total score'. The scores range between 0-100 where higher scores indicate a better quality of life. A positive change score indicates an improvement since baseline.
CagriSema 2.4 mg/2.4 mg versus placebo and semaglutide 2.4 mg: Number of Treatment Emergent Adverse Events (TEAEs) | From baseline (week 0) to end of study (week 51)
  Measured as count of events
CagriSema 2.4 mg/2.4 mg versus placebo and semaglutide 2.4 mg: Number of Treatment Emergent Serious Adverse Events (TESAEs) | From baseline (week 0) to end of study (week 51)
  Measured as count of events
Number of clinically significant hypoglycaemic episodes (level 2) (lesser than 3.0 mmol/L (54 milligrams per deciliter[mg/dL]), confirmed by BG meter) (only for participants with Type 2 diabetes (T2D) at screening) | From baseline (week 0) to end of study (week 51)
  Measured as count of episodes
Number of severe hypoglycaemic episodes (level 3): hypoglycaemia associated with severe cognitive impairment requiring external assistance for recovery, with no specific glucose threshold (only for participants with T2D at screening) | From baseline (week 0) to end of study (week 51)
  Measured as count of episodes

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Office (dept. 2834), Study Director — Novo Nordisk A/S
Locations (36):
- China (36):
  - Chinese People's Liberation Army General Hospital-Endocrinology, Beijing, Beijing Municipality
  - Chongqing University Three Gorges Hospital, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital-Endocrinology, Fuzhou, Fujian
  - Huizhou Central People's Hospital-Endocrinology, Huizhou, Guangdong
  - Hengshui People's Hospital (Harrison International Peace Hospital)-Endocrinology, Hengshui, Hebei
  - The Second Hospital of Hebei Medical University-Endocrinology, Shijiazhuang, Hebei
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Huaihe Hospital of Henan University-Endocrinology, Kaifeng, Henan
  - Huaihe Hospital of Henan University, Kaifeng, Henan
  - The First Affiliated Hospital of Henan University of Science and Technology-Endocrinology, Luoyang, Henan
  - The First Affiliated Hospital of Henan university of Science, Luoyang, Henan
  - The Second Affiliated Hospital of Zhengzhou University-Endocrinology, Zhengzhou, Henan
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The First People's Hospital of Changde City-Endocrinology, Changde, Hunan
  - Changzhou No.2 People's Hospital, Changzhou, Jiangsu
  - The First People's Hospital of Changzhou, Changzhou, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Suzhou Municipal Hospital-Endocrinology, Suzhou, Jiangsu
  - The First Affiliated Hospital of Soochow University-Endocrinology, Suzhou, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - The Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - The first hospital of Jilin University, Changchun, Jilin
  - The First Bethune hospital of Jilin University-Endocrinology, Changchun, Jilin
  - Jinan Central Hospital, Ji'nan, Shandong
  - Jinan Central Hospital, Jin'an, Shandong
  - Jinan Central Hospital, Jinan, Shandong
  - Huashan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Tongren Hospital Shanghai Jiao Tong Univ. School of Medicine, Shanghai, Shanghai Municipality
  - Tongren Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Central Hospital of Minhang District, Shanghai-Endocrinology, Shanghai, Shanghai Municipality
  - Central Hospital of Minhang District-Endocrinology, Shanghai, Shanghai Municipality
  - Shanghai Pudong New Area People's Hospital-Endocrinology, Shanghai, Shanghai Municipality
  - General Hospital of Tianjin Medical University-Endocrinology, Tianjin, Tianjin Municipality
  - General Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - The Second Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - Huashan Hospital Fudan University, Jingan/Shanghai

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com